CLINICAL TRIAL: NCT04447417
Title: Open Label Exploratory Study to Evaluate the Effect of Dupilumab on Skin Barrier Function in Patients With Moderate to Severe Atopic Dermatitis
Brief Title: Dupilumab Skin Barrier Function Study in Atopic Dermatitis
Acronym: BALISTAD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LPS15991; U1111-1244-1409 (Other: UTN); 2020-000314-15 (EudraCT Number)
Record Dates: First submitted 2020-06-22; First posted 2020-06-25 (Actual); Results first posted 2022-07-22 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — dupilumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Healthy Volunteer (No Intervention): Healthy volunteers with age, gender, location of targeted skin lesion area and study site matched to a selected atopic dermatitis (AD) participants, received no treatment, but were monitored in similar way as like enrolled AD participants.
- Atopic Dermatitis Patients (Experimental): Participants with moderate to severe AD and aged 18 years and older received dupilumab 600 milligrams (mg) (loading dose) subcutaneous (SC) injection on Day 1, followed by dupilumab 300 mg SC injection every 2 weeks (Q2W) through Week 14 (i.e., at Day 15, 29, 43, 57 and 85).
  Participants aged greater than or equal to (>=) 12 to less than (<) 18 years received treatment based on their body weight: <60 kilograms (kg) and >=60 kg - received dupilumab 400 mg and 600 mg (loading dose) SC injection on Day 1, respectively, followed by dupilumab 200 mg and 300 mg SC injection Q2W through Week 14 (i.e., at Day 15, 29, 43, 57 and 85).
  Interventions: Drug: Dupilumab SAR231893

INTERVENTIONS:
Drug: Dupilumab SAR231893 — Pharmaceutical form:solution for injection Route of administration: subcutaneous
  Other Names: REGN668
  Arms: Atopic Dermatitis Patients

SUMMARY:
Primary Objective:

- Evaluate changes in skin barrier function with transepidermal water loss (TEWL) assessed after skin tape stripping (STS) in pre-defined lesional skin in participants with moderate to severe atopic dermatitis (AD) treated with dupilumab.

Secondary Objectives:

* Evaluate changes in skin barrier function with TEWL assessed after STS in pre-defined lesional and non-lesional skin in participants with moderate to severe AD treated with dupilumab in reference to normal skin of healthy volunteers.
* Evaluate time course of skin barrier function with TEWL assessed before and after STS in pre-defined lesional and non-lesional skin in participants with moderate to severe AD treated with dupilumab in reference to normal skin of healthy volunteers.

DETAILED DESCRIPTION:
The duration for each participant was a total of approximately 24 weeks.

ELIGIBILITY:
Inclusion criteria :

- Participant must be between 12 to 65 years of age (inclusive), at the time of signing the informed consent.

Atopic dermatitis participants:

* Male or female participants.
* Participants with AD diagnosis according to Hanifin and Rajka criteria at least 1 year before screening.
* Investigator Global Assessment score of >=3 at screening (on the 0-4 scale).
* Participants with moderate to severe atopic dermatitis that were eligible to be treated with dupilumab according to product monograph.
* Participants with AD must have had active lesions on the upper limbs or lower limbs, with severity for lesion erythema or edema/papulation >=2 at screening on the 0-3 scale of the individual signs score.
* Patients must have had a non-lesional (normal looking) skin area 4 centimeters from the edge of the lesional area.
* Were willing to refrain from applying any topical medication products on the target assessment areas (including lesional and non-lesional) throughout the study unless necessary to alleviate intolerable symptoms.
* Were willing to refrain taking showers or soaking in a bathtub with soaps and body washes within 6 hours before TEWL assessments.
* Were willing to apply Cetaphil or Vanicream moisturizer up to twice a day with an exception of moisturizer application on the targeted assessment areas (lesional and non-lesional areas) during the entire study from Day -7 to end of treatment.
* Were willing and able to comply with all clinic visits and study-related procedures.

Healthy volunteers:

* Age and gender matched to a selected AD participant. Adolescents aged 12 to 17 years matched by post puberty status, and adults aged 18 to 65 years were matched by age as close as possible within 10 years of age.
* No current dermatologic or systemic condition that could interfere with the assessments.
* Contraceptive use by women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* Capable of understanding and giving signed informed consent/assent as were described in the protocol, which included compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. For adolescents >=12 and <18 years of age a specific ICF must also be signed by the participant's legally authorized representative.

Exclusion criteria:

* Skin conditions other than AD that can confound assessments in the area of TEWL assessments in the opinion of the investigator (i.e., skin atrophy, ichthyosis, Netherton syndrome, severe photo damage).
* Cracked, crusted, oozing, or bleeding AD lesions in the designated lesional assessment area leaving insufficient skin that was adequate for TEWL assessments.
* Hypersensitivity to the active substance or to any of the excipients of dupilumab.
* Ocular disorder that in the opinion of the investigator could adversely affect the individual's risk for study participation. Examples include -but are not limited to- individuals with a history of active cases of herpes keratitis; Sjogren's syndrome, keratoconjunctivitis sicca or dry eye syndrome that required daily use of supplemental lubrication; or individuals with ocular conditions that required the use of ocular corticosteroids or cyclosporine.
* Systemic AD treatment or phototherapy within 4 weeks of Baseline.
* Topical AD treatment within 1 week of Baseline. Face and neck may be treated with topical steroids during the washout period if approved by the investigator.
* Severe concomitant illness(es) that, in the investigator's judgment, would adversely affect the participant's participation in the study. Examples included, but were not limited to participants with short life expectancy, participants with uncontrolled diabetes (hemoglobin A1c >=9%), participants with cardiovascular conditions (eg, Class III or IV cardiac failure according to the New York Heart Association classification), severe renal conditions (eg, participants on dialysis), hepato-biliary conditions (eg, Child-Pugh class B or C), neurological conditions (eg, demyelinating diseases), active major autoimmune diseases (eg, lupus, inflammatory bowel disease, rheumatoid arthritis, etc.), other severe endocrinological, gastrointestinal, metabolic, pulmonary, psychiatric (known suicidal intentions) or lymphatic diseases. The specific justification for participants excluded under this criterion were noted in study documents (chart notes, electronic case report forms, screening logs, etc.).
* History of hypersensitivity reaction to tape or adhesives.
* Treatment with an investigational drug within 8 weeks or within 5 half-lives (if known) prior to Day 1, whichever was longer.
* Current participation in another investigational clinical study.
* Individuals accommodated in an institution because of regulatory or legal order; prisoners or participants who were legally institutionalized.
* Participants were dependent on the Sponsor or Investigator (in conjunction with section 1.61 of the ICH-GCP Ordinance E6).
* Individuals directly involved in the conduct of the study, or immediate family members of such individuals.
* Any specific situation during study implementation/course that might rise ethics considerations.
* Planned or anticipated major surgical procedure during the participant's participation in this study.
* Pregnant or breast feeding women, or were planning to become pregnant or breastfeed during the participant's participation in this study.
* Women unwilling to use adequate birth control, if of reproductive potential* and sexually active. Adequate birth control was defined as agreement to consistently practice an effective and accepted method of contraception throughout the duration of the study and for 12 weeks after last dose of study drug. These included condom, spermicide, hormonal contraceptives, intrauterine device, or double barrier contraception (i.e., condom + diaphragm) or a male partner with documented vasectomy. Additional requirements for acceptable contraception might apply in certain countries, based on local regulations. Investigators in these countries were notified accordingly in a protocol clarification letter.

  *For females, menopause was defined as at least 12 consecutive months without menses; if in question, a follicle stimulating hormone level of >=25 milliunits per milliliter must be documented. Hysterectomy, bilateral oophorectomy, or bilateral tubal ligation must be documented, as applicable; if documented, women with these conditions were not required to use additional contraception.
* Healthy volunteers with a personal history of an atopic condition.
* Healthy volunteers with use of any topical treatment anywhere except Cetaphil or Vanicream moisturizer on non-targeted skin areas.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2020-07-16 (Actual); Primary Completion 2021-06-17 (Actual); Study Completion 2021-06-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (2):
- Investigational Site Number 8400001, Denver, Colorado, United States
- Investigational Site Number 1240001, Montreal, Canada

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org.

REFERENCES:
- See also: LPS15991 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25277&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at 2 centers in the United States and Canada. A total of 52 eligible participants were enrolled between 16 July 2020 and 19 January 2021 under the AD participants cohort or the healthy volunteers cohort.
Pre-assignment Details: Healthy volunteer's cohort received no treatment and was considered as a reference comparator group.
Groups:
- Healthy Volunteer: Healthy volunteers with age, gender, location of targeted skin lesion area and study site matched to a selected atopic dermatitis (AD) participants, received no treatment, but were monitored in similar way as AD participants.
Period: Overall Study
Arm/Group | Healthy Volunteer | Atopic Dermatitis Patients
Started | 26 | 26
Completed | 23 | 26
Not Completed | 3 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Failure to meet inclusion criteria | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on safety population: all enrolled participants who actually received at least one dose of investigational medicinal product (IMP) or had at least one transepidermal water loss (TEWL)/skin tape stripping (STS) assessment and all healthy volunteers who had at least one TEWL/STS assessment performed.
Arm/Group | Healthy Volunteer | Atopic Dermatitis Patients | Total Title
Number analyzed (Participants) | 26 | 26 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.4 (16.4) | 32.2 (17.2) | 32.8 (16.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 15 | 15 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 21 | 21 | 42
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Transepidermal Water Loss After 5 Skin Tape Stripping (STS) on Lesional Skin (LS) in AD Patients at Week 16
Description: TEWL assessment: a noninvasive in vivo measurement of water loss across stratum corneum that is used to characterize skin barrier function (SBF). TEWL combined with STS measures SBF. With STS, the uppermost layers of the skin are peeled away using adhesive discs. Lesional skin (LS) areas for TEWL assessment and STS was identified at Baseline ('predefined skin area'). Within the predefined LS areas, 3 closely adjacent non-overlapping spots identified for subsequent SBF assessment. TEWL was measured prior to STS and after 5, 10, 15 and 20 STS on pre-defined LS areas at specified time points. STS assessment at Baseline (Week 0, Day 1) and Week 16 was conducted on first spot. Percent Change from Baseline at Week 16 in TEWL after 5 STS on LS (first spot) in AD participants were reported in this outcome measure (OM). Here, overall number of participants analyzed=participants evaluable for this OM.
Time Frame: Baseline, Week 16
Population: Modified intent-to-treat (mITT) population: all enrolled AD participants who received at least 1 dose of investigational medicinal product (IMP) and all enrolled healthy volunteers who had at least 1 TEWL/STS assessment performed, irrespective of compliance with protocol and procedures. If prohibited therapies used for AD, only visits prior to rescue treatment were considered. Data for this OM was not planned to be collected and analyzed for Healthy Volunteer arm as pre-specified in protocol.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Atopic Dermatitis Patients
Number analyzed (Participants) | 21
percent change | -54.6 (18.0)
Statistical Analysis 1: Comparison: Atopic Dermatitis Patients; TEWL data for linear mixed model was log-transformed to account for right skewness of data and heteroskedasticity. The linear mixed effect on log (TEWL) included age, sex, number of STS, localization on the body, visit, number of STS-by-visit interaction and number of STS-by-age interaction as fixed effects. Model was run on data on lesional skin area; Test type: Other; p <= 0.0001, linear mixed model — One-sided p-value. Threshold for significance at 0.05 level; Point estimate = 0.43, 90% CI 2-sided [0.37 to 0.49] — Point estimate obtained was back-transformed by exponentiation

2. Secondary Outcome: Percent Change From Baseline in TEWL After 20 STS on Lesional and Non-lesional Skin (Non-LS) in AD Patients at Week 16
Description: TEWL assessment: a noninvasive in vivo measurement of water loss across stratum corneum that is used to characterize SBF. TEWL combined with STS measures SBF. With STS, the uppermost layers of the skin are peeled away using adhesive discs. The LS and non-LS areas for TEWL assessment and STS were identified at Baseline ('predefined skin area'). Within the predefined LS and non-LS areas, 3 closely adjacent non-overlapping spots identified for subsequent SBF assessment (3 spots on LS, 3 spots on non-LS). TEWL was measured prior to STS and after 5, 10, 15 and 20 STS on pre-defined LS and non-LS areas at specified time points. STS assessment at Baseline (Week 0, Day 1) and Week 16 was conducted on first spot. Percent change from Baseline at Week 16 in TEWL after 20 STS on LS and non-LS (first spot) in AD participants were reported in this OM.
Time Frame: Baseline, Week 16
Population: Analysis was performed on mITT population. Here, number analyzed = participants with available data for each specified category. Data for this OM was not planned to be collected and analyzed for Healthy Volunteer arm as pre-specified in the protocol.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Atopic Dermatitis Patients
Number analyzed (Participants) | 26
percent change
  Lesional skin: number analyzed (Participants) | 7
  Lesional skin | -47.7 (20.1)
  Non-Lesional skin: number analyzed (Participants) | 21
  Non-Lesional skin | 16.6 (91.5)

3. Secondary Outcome: Absolute Change in TEWL After 20 STS on Lesional and Non-lesional Skin in AD Patients at Week 16
Description: TEWL assessment: a noninvasive in vivo measurement of water loss across stratum corneum that is used to characterize SBF. TEWL combined with STS measures SBF. With STS, the uppermost layers of the skin are peeled away using adhesive discs. The LS and non-LS areas for TEWL assessment and STS were identified at Baseline ('predefined skin area'). Within the predefined LS and non-LS areas, 3 closely adjacent non-overlapping spots identified for subsequent SBF assessment (3 spots on LS, 3 spots on non-LS). TEWL was measured prior to STS and after 5, 10, 15 and 20 STS on pre-defined LS and non-LS areas at specified time points. STS assessment at Baseline (Week 0, Day 1) and Week 16 was conducted on first spot. Absolute change from Baseline at Week 16 in TEWL after 20 STS on LS and non-LS (first spot) in AD participants were reported in this OM.
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: grams per square meter per hour
Arm/Group | Atopic Dermatitis Patients
Number analyzed (Participants) | 26
grams per square meter per hour
  Lesional skin: number analyzed (Participants) | 7
  Lesional skin | -42.6 (22.1)
  Non-Lesional skin: number analyzed (Participants) | 21
  Non-Lesional skin | -2.1 (26.2)

4. Secondary Outcome: Percent Change From Baseline in TEWL After 20 STS on Normal Skin in Healthy Volunteers at Week 16
Description: TEWL assessment: a noninvasive in vivo measurement of water loss across stratum corneum that is used to characterize SBF. TEWL combined with STS measures SBF. With STS, the uppermost layers of the skin are peeled away using adhesive discs. The normal skin areas for TEWL assessment and STS were identified at Baseline ('predefined skin area'). Within the predefined normal skin areas, 3 closely adjacent non-overlapping spots identified for subsequent SBF assessment. TEWL was measured prior to STS and after 5, 10, 15 and 20 STS on pre-defined normal skin areas at specified time points. STS assessment at Baseline (Week 0, Day 1) and Week 16 was conducted on first spot. Percent change from Baseline at Week 16 in TEWL after 20 STS on normal skin (first spot) in healthy volunteers were reported in this OM.
Time Frame: Baseline, Week 16
Population: Analysis was performed on mITT population. Here, overall number of participants analyzed = participants evaluable for this OM. Data for this OM was not planned to be collected and analyzed for Atopic Dermatitis Patients arm as pre-specified in the protocol.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Healthy Volunteer
Number analyzed (Participants) | 23
percent change | -5.8 (46.0)

5. Secondary Outcome: Absolute Change From Baseline in TEWL After 20 STS on Normal Skin in Healthy Volunteers at Week 16
Description: TEWL assessment: a noninvasive in vivo measurement of water loss across stratum corneum that is used to characterize SBF. TEWL combined with STS measures SBF. With STS, the uppermost layers of the skin are peeled away using adhesive discs. The normal skin areas for TEWL assessment and STS were identified at Baseline ('predefined skin area'). Within the predefined normal skin areas, 3 closely adjacent non-overlapping spots identified for subsequent SBF assessment. TEWL was measured prior to STS and after 5, 10, 15 and 20 STS on pre-defined normal skin areas at specified time points. STS assessment at Baseline (Week 0, Day 1) and Week 16 was conducted on first spot. Absolute change from Baseline at Week 16 in TEWL after 20 STS on normal skin (first spot) in healthy volunteers were reported in this OM.
Time Frame: Baseline, Week 16
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: grams per square meter per hour
Arm/Group | Healthy Volunteer
Number analyzed (Participants) | 23
grams per square meter per hour | -8.0 (19.2)

6. Secondary Outcome: Percent Change From Baseline in TEWL After 15 STS on Lesional and Non-lesional Skin in AD Patients at Week 16
Description: TEWL assessment: a noninvasive in vivo measurement of water loss across stratum corneum that is used to characterize SBF. TEWL combined with STS measures SBF. With STS, the uppermost layers of the skin are peeled away using adhesive discs. The LS and non-LS areas for TEWL assessment and STS were identified at Baseline ('predefined skin area'). Within the predefined LS and non-LS areas, 3 closely adjacent non-overlapping spots identified for subsequent SBF assessment (3 spots on LS, 3 spots on non-LS). TEWL was measured prior to STS and after 5, 10, 15 and 20 STS on pre-defined LS and non-LS areas at specified time points. STS assessment at Baseline (Week 0, Day 1) and Week 16 was conducted on first spot. Percent change from Baseline at Week 16 in TEWL after 15 STS on LS and non-LS (first spot) in AD participants were reported in this OM.
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Atopic Dermatitis Patients
Number analyzed (Participants) | 26
percent change
  Lesional skin: number analyzed (Participants) | 7
  Lesional skin | -51.2 (17.4)
  Non-Lesional skin: number analyzed (Participants) | 21
  Non-Lesional skin | 25.1 (116.5)

7. Secondary Outcome: Absolute Change From Baseline in TEWL After 15 STS on Lesional and Non-lesional Skin in AD Patients at Week 16
Description: TEWL assessment: a noninvasive in vivo measurement of water loss across stratum corneum that is used to characterize SBF. TEWL combined with STS measures SBF. With STS, the uppermost layers of the skin are peeled away using adhesive discs. The LS and non-LS areas for TEWL assessment and STS were identified at Baseline ('predefined skin area'). Within the predefined LS and non-LS areas, 3 closely adjacent non-overlapping spots identified for subsequent SBF assessment (3 spots on LS, 3 spots on non-LS). TEWL was measured prior to STS and after 5, 10, 15 and 20 STS on pre-defined LS and non-LS areas at specified time points. STS assessment at Baseline (Week 0, Day 1) and Week 16 was conducted on first spot. Absolute change from Baseline at Week 16 in TEWL after 15 STS on LS and non-LS (first spot) in AD participants were reported in this OM.
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: grams per square meter per hour
Arm/Group | Atopic Dermatitis Patients
Number analyzed (Participants) | 26
grams per square meter per hour
  Lesional skin: number analyzed (Participants) | 7
  Lesional skin | -43.1 (20.6)
  Non-Lesional skin: number analyzed (Participants) | 21
  Non-Lesional skin | -2.0 (23.5)

8. Secondary Outcome: Percent Change From Baseline in TEWL After 15 STS on Normal Skin in Healthy Volunteers at Week 16
Description: TEWL assessment: a noninvasive in vivo measurement of water loss across stratum corneum that is used to characterize SBF. TEWL combined with STS measures SBF. With STS, the uppermost layers of the skin are peeled away using adhesive discs. The normal skin areas for TEWL assessment and STS were identified at Baseline ('predefined skin area'). Within the predefined normal skin areas, 3 closely adjacent non-overlapping spots identified for subsequent SBF assessment. TEWL was measured prior to STS and after 5, 10, 15 and 20 STS on pre-defined normal skin areas at specified time points. STS assessment at Baseline (Week 0, Day 1) and Week 16 was conducted on first spot. Percent change from Baseline at Week 16 in TEWL after 15 STS on normal skin (first spot) in healthy volunteers were reported in this OM.
Time Frame: Baseline, Week 16
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Healthy Volunteer
Number analyzed (Participants) | 23
percent change | -7.2 (35.8)

9. Secondary Outcome: Absolute Change From Baseline in TEWL After 15 STS on Normal Skin in Healthy Volunteers at Week 16
Description: TEWL assessment: a noninvasive in vivo measurement of water loss across stratum corneum that is used to characterize SBF. TEWL combined with STS measures SBF. With STS, the uppermost layers of the skin are peeled away using adhesive discs. The normal skin areas for TEWL assessment and STS were identified at Baseline ('predefined skin area'). Within the predefined normal skin areas, 3 closely adjacent non-overlapping spots identified for subsequent SBF assessment. TEWL was measured prior to STS and after 5, 10, 15 and 20 STS on pre-defined normal skin areas at specified time points. STS assessment at Baseline (Week 0, Day 1) and Week 16 was conducted on first spot. Absolute change from Baseline at Week 16 in TEWL after 15 STS on normal skin (first spot) in healthy volunteers were reported in this OM.
Time Frame: Baseline, Week 16
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: grams per square meter per hour
Arm/Group | Healthy Volunteer
Number analyzed (Participants) | 23
grams per square meter per hour | -4.5 (11.1)

10. Secondary Outcome: Percent Change From Baseline in TEWL After 10 STS on Lesional and Non-lesional Skin in AD Patients at Week 16
Description: TEWL assessment: a noninvasive in vivo measurement of water loss across stratum corneum that is used to characterize SBF. TEWL combined with STS measures SBF. With STS, the uppermost layers of the skin are peeled away using adhesive discs. The LS and non-LS areas for TEWL assessment and STS were identified at Baseline ('predefined skin area'). Within the predefined LS and non-LS areas, 3 closely adjacent non-overlapping spots identified for subsequent SBF assessment (3 spots on LS, 3 spots on non-LS). TEWL was measured prior to STS and after 5, 10, 15 and 20 STS on pre-defined LS and non-LS areas at specified time points. STS assessment at Baseline (Week 0, Day 1) and Week 16 was conducted on first spot. Percent change from Baseline at Week 16 in TEWL after 10 STS on LS and non-LS (first spot) in AD participants were reported in this OM.
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Atopic Dermatitis Patients
Number analyzed (Participants) | 26
percent change
  Lesional skin: number analyzed (Participants) | 20
  Lesional skin | -54.9 (17.5)
  Non-Lesional skin: number analyzed (Participants) | 21
  Non-Lesional skin | 26.2 (111.8)

11. Secondary Outcome: Absolute Change From Baseline in TEWL After 10 STS on Lesional and Non-lesional Skin in AD Patients at Week 16
Description: TEWL assessment: a noninvasive in vivo measurement of water loss across stratum corneum that is used to characterize SBF. TEWL combined with STS measures SBF. With STS, the uppermost layers of the skin are peeled away using adhesive discs. The LS and non-LS areas for TEWL assessment and STS were identified at Baseline ('predefined skin area'). Within the predefined LS and non-LS areas, 3 closely adjacent non-overlapping spots identified for subsequent SBF assessment (3 spots on LS, 3 spots on non-LS). TEWL was measured prior to STS and after 5, 10, 15 and 20 STS on pre-defined LS and non-LS areas at specified time points. STS assessment at Baseline (Week 0, Day 1) and Week 16 was conducted on first spot. Absolute change from Baseline at Week 16 in TEWL after 10 STS on LS and non-LS (first spot) in AD participants were reported in this OM.
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: grams per square meter per hour
Arm/Group | Atopic Dermatitis Patients
Number analyzed (Participants) | 26
grams per square meter per hour
  Lesional skin: number analyzed (Participants) | 20
  Lesional skin | -41.2 (20.4)
  Non-Lesional skin: number analyzed (Participants) | 21
  Non-Lesional skin | -0.5 (17.9)

12. Secondary Outcome: Percent Change From Baseline in TEWL After 10 STS on Normal Skin in Healthy Volunteers at Week 16
Description: TEWL assessment: a noninvasive in vivo measurement of water loss across stratum corneum that is used to characterize SBF. TEWL combined with STS measures SBF. With STS, the uppermost layers of the skin are peeled away using adhesive discs. The normal skin areas for TEWL assessment and STS were identified at Baseline ('predefined skin area'). Within the predefined normal skin areas, 3 closely adjacent non-overlapping spots identified for subsequent SBF assessment. TEWL was measured prior to STS and after 5, 10, 15 and 20 STS on pre-defined normal skin areas at specified time points. STS assessment at Baseline (Week 0, Day 1) and Week 16 was conducted on first spot. Percent change from Baseline at Week 16 in TEWL after 10 STS on normal skin (first spot) in healthy volunteers were reported in this OM.
Time Frame: Baseline, Week 16
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Healthy Volunteer
Number analyzed (Participants) | 22
percent change | -2.0 (23.5)

13. Secondary Outcome: Absolute Change From Baseline in TEWL After 10 STS on Normal Skin in Healthy Volunteers at Week 16
Description: TEWL assessment: a noninvasive in vivo measurement of water loss across stratum corneum that is used to characterize SBF. TEWL combined with STS measures SBF. With STS, the uppermost layers of the skin are peeled away using adhesive discs. The normal skin areas for TEWL assessment and STS were identified at Baseline ('predefined skin area'). Within the predefined normal skin areas, 3 closely adjacent non-overlapping spots identified for subsequent SBF assessment. TEWL was measured prior to STS and after 5, 10, 15 and 20 STS on pre-defined normal skin areas at specified time points. STS assessment at Baseline (Week 0, Day 1) and Week 16 was conducted on first spot. Absolute change from Baseline at Week 16 in TEWL after 10 STS on normal skin (first spot) in healthy volunteers were reported in this OM.
Time Frame: Baseline, Week 16
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: grams per square meter per hour
Arm/Group | Healthy Volunteer
Number analyzed (Participants) | 22
grams per square meter per hour | -0.8 (4.0)

14. Secondary Outcome: Absolute Change From Baseline in TEWL After 5 STS on Lesional Skin in AD Patients at Week 16
Description: TEWL assessment: a noninvasive in vivo measurement of water loss across stratum corneum that is used to characterize SBF. TEWL combined with STS measures SBF. With STS, the uppermost layers of the skin are peeled away using adhesive discs. The LS areas for TEWL assessment and STS were identified at Baseline ('predefined skin area'). Within the predefined LS areas, 3 closely adjacent non-overlapping spots identified for subsequent SBF assessment. TEWL was measured prior to STS and after 5, 10, 15 and 20 STS on pre-defined LS areas at specified time points. STS assessment at Baseline (Week 0, Day 1) and Week 16 was conducted on first spot. Absolute change from Baseline at Week 16 in TEWL after 5 STS on LS (first spot) in AD participants were reported in this OM.
Time Frame: Baseline, Week 16
Population: Analysis was performed on mITT population. Here, overall number of participants analyzed = participants evaluable for this OM. Data for this OM was not planned to be collected and analyzed for Healthy Volunteer arm as pre-specified in the protocol.
Measure: Mean (Standard Deviation); unit: grams per square meter per hour
Arm/Group | Atopic Dermatitis Patients
Number analyzed (Participants) | 21
grams per square meter per hour | -35.1 (17.1)

15. Secondary Outcome: Percent Change From Baseline in TEWL After 5 STS on Non-lesional Skin in AD Patients at Week 16
Description: TEWL assessment: a noninvasive in vivo measurement of water loss across stratum corneum that is used to characterize SBF. TEWL combined with STS measures SBF. With STS, the uppermost layers of the skin are peeled away using adhesive discs. The non-LS areas for TEWL assessment and STS were identified at Baseline ('predefined skin area'). Within the predefined non-LS areas, 3 closely adjacent non-overlapping spots identified for subsequent SBF assessment. TEWL was measured prior to STS and after 5, 10, 15 and 20 STS on pre-defined non-LS areas at specified time points. STS assessment at Baseline (Week 0, Day 1) and Week 16 was conducted on first spot. Percent change from Baseline at Week 16 in TEWL after 5 STS on non-LS (first spot) in AD participants were reported in this OM.
Time Frame: Baseline, Week 16
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Atopic Dermatitis Patients
Number analyzed (Participants) | 20
percent change | 17.6 (82.2)

16. Secondary Outcome: Absolute Change From Baseline in TEWL After 5 STS on Non-lesional Skin in AD Patients at Week 16
Description: TEWL assessment: a noninvasive in vivo measurement of water loss across stratum corneum that is used to characterize SBF. TEWL combined with STS measures SBF. With STS, the uppermost layers of the skin are peeled away using adhesive discs. The non-LS areas for TEWL assessment and STS were identified at Baseline ('predefined skin area'). Within the predefined non-LS areas, 3 closely adjacent non-overlapping spots identified for subsequent SBF assessment. TEWL was measured prior to STS and after 5, 10, 15 and 20 STS on pre-defined non-LS areas at specified time points. STS assessment at Baseline (Week 0, Day 1) and Week 16 was conducted on first spot. Absolute change from Baseline at Week 16 in TEWL after 5 STS on non-LS (first spot) in AD participants were reported in this OM.
Time Frame: Baseline, Week 16
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: grams per square meter per hour
Arm/Group | Atopic Dermatitis Patients
Number analyzed (Participants) | 20
grams per square meter per hour | -0.8 (13.6)

17. Secondary Outcome: Percent Change From Baseline in TEWL After 5 STS on Normal Skin in Healthy Volunteers at Week 16
Description: TEWL assessment: a noninvasive in vivo measurement of water loss across stratum corneum that is used to characterize SBF. TEWL combined with STS measures SBF. With STS, the uppermost layers of the skin are peeled away using adhesive discs. The normal skin areas for TEWL assessment and STS were identified at Baseline ('predefined skin area'). Within the predefined normal skin areas, 3 closely adjacent non-overlapping spots identified for subsequent SBF assessment. TEWL was measured prior to STS and after 5, 10, 15 and 20 STS on pre-defined normal skin areas at specified time points. STS assessment at Baseline (Week 0, Day 1) and Week 16 was conducted on first spot. Percent change from Baseline at Week 16 in TEWL after 5 STS on normal skin (first spot) in healthy volunteers were reported in this OM.
Time Frame: Baseline, Week 16
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Healthy Volunteer
Number analyzed (Participants) | 23
percent change | 1.2 (21.9)

18. Secondary Outcome: Absolute Change From Baseline in TEWL After 5 STS on Normal Skin in Healthy Volunteers at Week 16
Description: TEWL assessment: a noninvasive in vivo measurement of water loss across stratum corneum that is used to characterize SBF. TEWL combined with STS measures SBF. With STS, the uppermost layers of the skin are peeled away using adhesive discs. The normal skin areas for TEWL assessment and STS were identified at Baseline ('predefined skin area'). Within the predefined normal skin areas, 3 closely adjacent non-overlapping spots identified for subsequent SBF assessment. TEWL was measured prior to STS and after 5, 10, 15 and 20 STS on pre-defined normal skin areas at specified time points. STS assessment at Baseline (Week 0, Day 1) and Week 16 was conducted on first spot. Absolute change from Baseline at Week 16 in TEWL after 5 STS on normal skin (first spot) in healthy volunteers were reported in this OM.
Time Frame: Baseline, Week 16
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: grams per square meter per hour
Arm/Group | Healthy Volunteer
Number analyzed (Participants) | 23
grams per square meter per hour | 0.0 (2.7)

19. Secondary Outcome: Percent Change From Baseline in TEWL Before STS on Lesional and Non-lesional Skin in AD Patients at Day 4, 8, 11, 15, 22, 29, 43, 57, 85 and Week 16
Description: TEWL assessment: a noninvasive in vivo measurement of water loss across stratum corneum that is used to characterize SBF. LS and non-LS areas for TEWL assessment were identified at Baseline ('predefined skin area'). Within predefined LS and non-LS areas, 3 closely adjacent non-overlapping spots identified for subsequent SBF assessment (3 spots on LS, 3 spots on non-LS). TEWL was measured prior to STS on pre-defined LS and non-LS areas at specified time points. At each visit, before STS, all three spots were assessed, and their value was averaged to derive a single value. Percent change from Baseline at specified time points in TEWL before STS on LS and non-LS in AD participants were reported in this OM.
Time Frame: Baseline, Day 4, 8, 11, 15, 22, 29, 43, 57, 85 and Week 16
Population: Analyzed on mITT population. Here, number analyzed = participants with available data for each specified category. Data for this OM was not planned to be collected and analyzed for Healthy Volunteer arm as pre-specified in the protocol.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Atopic Dermatitis Patients
Number analyzed (Participants) | 26
percent change
  Lesional skin: Day 4: number analyzed (Participants) | 24
  Lesional skin: Day 4 | -0.7 (30.1)
  Lesional skin: Day 8: number analyzed (Participants) | 25
  Lesional skin: Day 8 | -5.3 (42.1)
  Lesional skin: Day 11: number analyzed (Participants) | 24
  Lesional skin: Day 11 | -12.9 (32.6)
  Lesional skin: Day 15: number analyzed (Participants) | 25
  Lesional skin: Day 15 | -16.3 (34.5)
  Lesional skin: Day 22: number analyzed (Participants) | 25
  Lesional skin: Day 22 | -37.8 (20.6)
  Lesional skin: Day 29: number analyzed (Participants) | 24
  Lesional skin: Day 29 | -35.1 (19.9)
  Lesional skin: Day 43: number analyzed (Participants) | 23
  Lesional skin: Day 43 | -40.6 (21.4)
  Lesional skin: Day 57: number analyzed (Participants) | 23
  Lesional skin: Day 57 | -42.1 (20.9)
  Lesional skin: Day 85: number analyzed (Participants) | 21
  Lesional skin: Day 85 | -42.7 (23.8)
  Lesional skin: Week 16: number analyzed (Participants) | 21
  Lesional skin: Week 16 | -48.7 (22.6)
  Non-Lesional skin: Day 4: number analyzed (Participants) | 24
  Non-Lesional skin: Day 4 | 25.2 (40.6)
  Non-Lesional skin: Day 8: number analyzed (Participants) | 25
  Non-Lesional skin: Day 8 | 27.9 (59.5)
  Non-Lesional skin: Day 11: number analyzed (Participants) | 24
  Non-Lesional skin: Day 11 | 20.1 (46.8)
  Non-Lesional skin: Day 15: number analyzed (Participants) | 25
  Non-Lesional skin: Day 15 | 24.0 (56.1)
  Non-Lesional skin: Day 22: number analyzed (Participants) | 25
  Non-Lesional skin: Day 22 | 14.5 (47.8)
  Non-Lesional skin: Day 29: number analyzed (Participants) | 24
  Non-Lesional skin: Day 29 | 6.4 (47.0)
  Non-Lesional skin: Day 43: number analyzed (Participants) | 23
  Non-Lesional skin: Day 43 | 5.6 (57.2)
  Non-Lesional skin: Day 57: number analyzed (Participants) | 23
  Non-Lesional skin: Day 57 | 17.8 (85.4)
  Non-Lesional skin: Day 85: number analyzed (Participants) | 21
  Non-Lesional skin: Day 85 | 27.5 (99.1)
  Non-Lesional skin: Week 16: number analyzed (Participants) | 21
  Non-Lesional skin: Week 16 | 18.8 (85.2)

20. Secondary Outcome: Absolute Change From Baseline up to Week 16 in TEWL Before STS on Lesional and Non-lesional Skin in AD Patients at Day 4, 8, 11, 15, 22, 29, 43, 57, 85 and Week 16
Description: TEWL assessment: noninvasive in vivo measurement of water loss across stratum corneum that is used to characterize SBF. LS and non-LS areas for TEWL assessment were identified at Baseline ('predefined skin area'). Within predefined LS and non-LS areas, 3 closely adjacent non-overlapping spots identified for subsequent SBF assessment (3 spots on LS, 3 spots on non-LS). TEWL was measured prior to STS on pre-defined LS and non-LS areas at specified time points. At each visit, before STS, all three spots were assessed, and their value was averaged to derive a single value. Absolute change from Baseline at specified time points in TEWL before STS on LS and non-LS in AD participants were reported in this OM.
Time Frame: Baseline, Day 4, 8, 11, 15, 22, 29, 43, 57, 85 and Week 16
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: grams per square meter per hour
Arm/Group | Atopic Dermatitis Patients
Number analyzed (Participants) | 26
grams per square meter per hour
  Lesional skin: Day 4: number analyzed (Participants) | 24
  Lesional skin: Day 4 | -3.0 (14.0)
  Lesional skin: Day 8: number analyzed (Participants) | 25
  Lesional skin: Day 8 | -5.6 (18.8)
  Lesional skin: Day 11: number analyzed (Participants) | 24
  Lesional skin: Day 11 | -8.2 (16.0)
  Lesional skin: Day 15: number analyzed (Participants) | 25
  Lesional skin: Day 15 | -10.4 (16.6)
  Lesional skin: Day 22: number analyzed (Participants) | 25
  Lesional skin: Day 22 | -19.3 (14.0)
  Lesional skin: Day 29: number analyzed (Participants) | 24
  Lesional skin: Day 29 | -17.7 (14.4)
  Lesional skin: Day 43: number analyzed (Participants) | 23
  Lesional skin: Day 43 | -20.9 (14.9)
  Lesional skin: Day 57: number analyzed (Participants) | 23
  Lesional skin: Day 57 | -20.9 (14.0)
  Lesional skin: Day 85: number analyzed (Participants) | 21
  Lesional skin: Day 85 | -22.4 (16.7)
  Lesional skin: Week 16: number analyzed (Participants) | 21
  Lesional skin: Week 16 | -24.3 (16.3)
  Non-Lesional skin: Day 4: number analyzed (Participants) | 24
  Non-Lesional skin: Day 4 | 2.7 (7.6)
  Non-Lesional skin: Day 8: number analyzed (Participants) | 25
  Non-Lesional skin: Day 8 | 3.8 (11.0)
  Non-Lesional skin: Day 11: number analyzed (Participants) | 24
  Non-Lesional skin: Day 11 | 2.1 (10.1)
  Non-Lesional skin: Day 15: number analyzed (Participants) | 25
  Non-Lesional skin: Day 15 | 2.6 (11.5)
  Non-Lesional skin: Day 22: number analyzed (Participants) | 25
  Non-Lesional skin: Day 22 | 0.4 (8.9)
  Non-Lesional skin: Day 29: number analyzed (Participants) | 24
  Non-Lesional skin: Day 29 | -1.2 (11.1)
  Non-Lesional skin: Day 43: number analyzed (Participants) | 23
  Non-Lesional skin: Day 43 | -1.7 (9.4)
  Non-Lesional skin: Day 57: number analyzed (Participants) | 23
  Non-Lesional skin: Day 57 | -0.9 (13.0)
  Non-Lesional skin: Day 85: number analyzed (Participants) | 21
  Non-Lesional skin: Day 85 | 1.0 (15.3)
  Non-Lesional skin: Week 16: number analyzed (Participants) | 21
  Non-Lesional skin: Week 16 | -0.7 (12.3)

21. Secondary Outcome: Percent Change From Baseline in TEWL Before STS on Normal Skin in Healthy Volunteers at Day 4, 8, 11, 15, 22, 29, 43, 57, 85 and Week 16
Description: TEWL assessment: noninvasive in vivo measurement of water loss across stratum corneum that is used to characterize SBF. Normal skin areas for TEWL assessment were identified at Baseline ('predefined skin area'). Within predefined normal skin areas, 3 closely adjacent non-overlapping spots identified for subsequent SBF assessment. TEWL was measured prior to STS on pre-defined normal skin areas at specified time points. At each visit, before STS, all three spots were assessed, and their value was averaged to derive a single value. Percent change from Baseline at specified time points in TEWL before STS on normal skin in healthy volunteers were reported in this OM.
Time Frame: Baseline, Day 4, 8, 11, 15, 22, 29, 43, 57, 85 and Week 16
Population: Analyzed on mITT population. Here, overall number of participants analyzed = participants evaluable for this OM and number analyzed = participants with available data for each specified category. Data for this OM was not planned to be collected and analyzed for Atopic Dermatitis Patients arm as pre-specified in the protocol.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Healthy Volunteer
Number analyzed (Participants) | 24
percent change
  Day 4 | 42.6 (44.4)
  Day 8: number analyzed (Participants) | 23
  Day 8 | 20.5 (38.4)
  Day 11: number analyzed (Participants) | 23
  Day 11 | 15.9 (31.0)
  Day 15: number analyzed (Participants) | 23
  Day 15 | 16.6 (25.1)
  Day 22: number analyzed (Participants) | 23
  Day 22 | 18.5 (32.2)
  Day 29: number analyzed (Participants) | 23
  Day 29 | 8.0 (20.2)
  Day 43: number analyzed (Participants) | 23
  Day 43 | 4.0 (26.2)
  Day 57: number analyzed (Participants) | 23
  Day 57 | 20.3 (31.9)
  Day 85: number analyzed (Participants) | 23
  Day 85 | 6.0 (21.8)
  Week 16: number analyzed (Participants) | 23
  Week 16 | 4.3 (25.3)

22. Secondary Outcome: Absolute Change From Baseline in TEWL Before STS on Normal Skin in Healthy Volunteers at Day 4, 8, 11, 15, 22, 29, 43, 57, 85 and Week 16
Description: TEWL assessment: noninvasive in vivo measurement of water loss across stratum corneum that is used to characterize SBF. Normal skin areas for TEWL assessment were identified at Baseline ('predefined skin area'). Within predefined normal skin areas, 3 closely adjacent non-overlapping spots identified for subsequent SBF assessment. TEWL was measured prior to STS on pre-defined normal skin areas at specified time points. At each visit, before STS, all three spots were assessed, and their value was averaged to derive a single value. Absolute change from Baseline at specified time points in TEWL before STS on normal skin in healthy volunteers were reported in this OM.
Time Frame: Baseline, Day 4, 8, 11, 15, 22, 29, 43, 57, 85 and Week 16
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: grams per square meter per hour
Arm/Group | Healthy Volunteer
Number analyzed (Participants) | 24
grams per square meter per hour
  Day 4 | 3.9 (4.6)
  Day 8: number analyzed (Participants) | 23
  Day 8 | 1.4 (3.1)
  Day 11: number analyzed (Participants) | 23
  Day 11 | 1.2 (3.3)
  Day 15: number analyzed (Participants) | 23
  Day 15 | 1.5 (2.7)
  Day 22: number analyzed (Participants) | 23
  Day 22 | 1.4 (2.5)
  Day 29: number analyzed (Participants) | 23
  Day 29 | 0.4 (2.2)
  Day 43: number analyzed (Participants) | 23
  Day 43 | -0.1 (2.7)
  Day 57: number analyzed (Participants) | 23
  Day 57 | 1.6 (4.0)
  Day 85: number analyzed (Participants) | 23
  Day 85 | 0.1 (2.7)
  Week 16: number analyzed (Participants) | 23
  Week 16 | 0.4 (2.8)

23. Secondary Outcome: Percent Change From Baseline in TEWL After 5, 10, 15 and 20 STS on Lesional and Non-lesional Skin in AD Patients at Day 15, 29, 57, 85 and Week 16
Description: TEWL assessment: noninvasive in vivo measurement of water loss across stratum corneum that is used to characterize SBF. TEWL combined with STS measures SBF. With STS, uppermost layers of skin are peeled away using adhesive discs. LS and non-LS areas for TEWL assessment and STS were identified at Baseline ('predefined skin area'). Within predefined LS and non-LS areas, 3 closely adjacent non-overlapping spots identified for subsequent SBF assessment (3 spots on LS, 3 spots on non-LS). TEWL: measured prior to STS and after 5, 10, 15 and 20 STS on pre-defined LS and non-LS areas at specified time points. STS assessment was done at Baseline (Week 0, Day 1), Day 57 and Week 16 on 1st spot; at Day 15 on 2nd spot and at Day 29 and Day 85 on 3rd spot. Percent change from Baseline at specified time points in TEWL after STS on LS and non-LS in AD participants were reported in this OM.
Time Frame: Baseline, Day 15, 29, 57, 85 and Week 16
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Atopic Dermatitis Patients
Number analyzed (Participants) | 26
percent change
  Lesional skin: After 5 STS: Day 15: number analyzed (Participants) | 25
  Lesional skin: After 5 STS: Day 15 | -25.1 (34.0)
  Lesional skin: After 5 STS: Day 29: number analyzed (Participants) | 24
  Lesional skin: After 5 STS: Day 29 | -38.9 (23.4)
  Lesional skin: After 5 STS: Day 57: number analyzed (Participants) | 23
  Lesional skin: After 5 STS: Day 57 | -45.6 (23.5)
  Lesional skin: After 5 STS: Day 85: number analyzed (Participants) | 20
  Lesional skin: After 5 STS: Day 85 | -50.6 (26.7)
  Lesional skin: After 5 STS: Week 16: number analyzed (Participants) | 21
  Lesional skin: After 5 STS: Week 16 | -54.6 (18.0)
  Lesional skin: After 10 STS: Day 15: number analyzed (Participants) | 24
  Lesional skin: After 10 STS: Day 15 | -18.5 (30.7)
  Lesional skin: After 10 STS: Day 29: number analyzed (Participants) | 24
  Lesional skin: After 10 STS: Day 29 | -32.5 (29.1)
  Lesional skin: After 10 STS: Day 57: number analyzed (Participants) | 23
  Lesional skin: After 10 STS: Day 57 | -46.7 (22.4)
  Lesional skin: After 10 STS: Day 85: number analyzed (Participants) | 21
  Lesional skin: After 10 STS: Day 85 | -47.0 (25.6)
  Lesional skin: After 10 STS: Week 16: number analyzed (Participants) | 20
  Lesional skin: After 10 STS: Week 16 | -54.9 (17.5)
  Lesional skin: After 15 STS: Day 15: number analyzed (Participants) | 9
  Lesional skin: After 15 STS: Day 15 | -14.5 (24.8)
  Lesional skin: After 15 STS: Day 29: number analyzed (Participants) | 10
  Lesional skin: After 15 STS: Day 29 | -33.0 (17.7)
  Lesional skin: After 15 STS: Day 57: number analyzed (Participants) | 8
  Lesional skin: After 15 STS: Day 57 | -39.1 (22.3)
  Lesional skin: After 15 STS: Day 85: number analyzed (Participants) | 7
  Lesional skin: After 15 STS: Day 85 | -43.4 (24.4)
  Lesional skin: After 15 STS: Week 16: number analyzed (Participants) | 7
  Lesional skin: After 15 STS: Week 16 | -51.2 (17.4)
  Lesional skin: After 20 STS: Day 15: number analyzed (Participants) | 9
  Lesional skin: After 20 STS: Day 15 | -11.6 (27.9)
  Lesional skin: After 20 STS: Day 29: number analyzed (Participants) | 10
  Lesional skin: After 20 STS: Day 29 | -29.1 (18.8)
  Lesional skin: After 20 STS: Day 57: number analyzed (Participants) | 9
  Lesional skin: After 20 STS: Day 57 | -37.4 (22.9)
  Lesional skin: After 20 STS: Day 85: number analyzed (Participants) | 7
  Lesional skin: After 20 STS: Day 85 | -38.8 (28.2)
  Lesional skin: After 20 STS: Week 16: number analyzed (Participants) | 7
  Lesional skin: After 20 STS: Week 16 | -47.7 (20.1)
  Non-Lesional skin: After 5 STS: Day 15: number analyzed (Participants) | 24
  Non-Lesional skin: After 5 STS: Day 15 | 49.8 (100.0)
  Non-Lesional skin: After 5 STS: Day 29: number analyzed (Participants) | 23
  Non-Lesional skin: After 5 STS: Day 29 | 8.0 (46.1)
  Non-Lesional skin: After 5 STS: Day 57: number analyzed (Participants) | 22
  Non-Lesional skin: After 5 STS: Day 57 | 22.8 (89.0)
  Non-Lesional skin: After 5 STS: Day 85: number analyzed (Participants) | 20
  Non-Lesional skin: After 5 STS: Day 85 | 33.7 (106.8)
  Non-Lesional skin: After 5 STS: Week 16: number analyzed (Participants) | 20
  Non-Lesional skin: After 5 STS: Week 16 | 17.6 (82.2)
  Non-Lesional skin: After 10 STS: Day 15: number analyzed (Participants) | 25
  Non-Lesional skin: After 10 STS: Day 15 | 55.1 (109.3)
  Non-Lesional skin: After 10 STS: Day 29: number analyzed (Participants) | 24
  Non-Lesional skin: After 10 STS: Day 29 | 4.5 (52.9)
  Non-Lesional skin: After 10 STS: Day 57: number analyzed (Participants) | 23
  Non-Lesional skin: After 10 STS: Day 57 | 18.6 (91.0)
  Non-Lesional skin: After 10 STS: Day 85: number analyzed (Participants) | 21
  Non-Lesional skin: After 10 STS: Day 85 | 31.0 (116.3)
  Non-Lesional skin: After 10 STS: Week 16: number analyzed (Participants) | 21
  Non-Lesional skin: After 10 STS: Week 16 | 26.2 (111.8)
  Non-Lesional skin: After 15 STS: Day 15: number analyzed (Participants) | 25
  Non-Lesional skin: After 15 STS: Day 15 | 70.9 (128.3)
  Non-Lesional skin: After 15 STS: Day 29: number analyzed (Participants) | 24
  Non-Lesional skin: After 15 STS: Day 29 | 2.4 (58.9)
  Non-Lesional skin: After 15 STS: Day 57: number analyzed (Participants) | 23
  Non-Lesional skin: After 15 STS: Day 57 | 23.5 (104.4)
  Non-Lesional skin: After 15 STS: Day 85: number analyzed (Participants) | 21
  Non-Lesional skin: After 15 STS: Day 85 | 34.7 (112.0)
  Non-Lesional skin: After 15 STS: Week 16: number analyzed (Participants) | 21
  Non-Lesional skin: After 15 STS: Week 16 | 25.1 (116.5)
  Non-Lesional skin: After 20 STS: Day 15: number analyzed (Participants) | 25
  Non-Lesional skin: After 20 STS: Day 15 | 53.1 (96.0)
  Non-Lesional skin: After 20 STS: Day 29: number analyzed (Participants) | 24
  Non-Lesional skin: After 20 STS: Day 29 | -3.8 (53.2)
  Non-Lesional skin: After 20 STS: Day 57: number analyzed (Participants) | 23
  Non-Lesional skin: After 20 STS: Day 57 | 14.3 (80.7)
  Non-Lesional skin: After 20 STS: Day 85: number analyzed (Participants) | 21
  Non-Lesional skin: After 20 STS: Day 85 | 30.4 (104.9)
  Non-Lesional skin: After 20 STS: Week 16: number analyzed (Participants) | 21
  Non-Lesional skin: After 20 STS: Week 16 | 16.6 (91.5)

24. Secondary Outcome: Absolute Change From Baseline in TEWL After 5, 10, 15 and 20 STS on Lesional and Non-lesional Skin in AD Patients at Day 15, 29, 57, 85 and Week 16
Description: TEWL assessment: noninvasive in vivo measurement of water loss across stratum corneum that is used to characterize SBF. TEWL combined with STS measures SBF. With STS, uppermost layers of skin are peeled away using adhesive discs. LS and non-LS areas for TEWL assessment and STS were identified at Baseline ('predefined skin area'). Within predefined LS and non-LS areas, 3 closely adjacent non-overlapping spots identified for subsequent SBF assessment (3 spots on LS, 3 spots on non-LS). TEWL: measured prior to STS and after 5, 10, 15 and 20 STS on pre-defined LS and non-LS areas at specified time points. STS assessment was done at Baseline (Week 0, Day 1), Day 57 and Week 16 on 1st spot; at Day 15 on 2nd spot and at Day 29 and Day 85 on 3rd spot. Absolute change from Baseline at specified time points in TEWL after STS on LS and non-LS in AD participants were reported in this OM.
Time Frame: Baseline, Day 15, 29, 57, 85 and Week 16
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: grams per square meter per hour
Arm/Group | Atopic Dermatitis Patients
Number analyzed (Participants) | 26
grams per square meter per hour
  Lesional skin: After 5 STS: Day 15: number analyzed (Participants) | 25
  Lesional skin: After 5 STS: Day 15 | -19.4 (21.8)
  Lesional skin: After 5 STS: Day 29: number analyzed (Participants) | 24
  Lesional skin: After 5 STS: Day 29 | -27.1 (20.2)
  Lesional skin: After 5 STS: Day 57: number analyzed (Participants) | 23
  Lesional skin: After 5 STS: Day 57 | -29.4 (19.1)
  Lesional skin: After 5 STS: Day 85: number analyzed (Participants) | 20
  Lesional skin: After 5 STS: Day 85 | -34.8 (21.6)
  Lesional skin: After 5 STS: Week 16: number analyzed (Participants) | 21
  Lesional skin: After 5 STS: Week 16 | -35.1 (17.1)
  Lesional skin: After 10 STS: Day 15: number analyzed (Participants) | 24
  Lesional skin: After 10 STS: Day 15 | -17.7 (24.5)
  Lesional skin: After 10 STS: Day 29: number analyzed (Participants) | 24
  Lesional skin: After 10 STS: Day 29 | -28.3 (25.9)
  Lesional skin: After 10 STS: Day 57: number analyzed (Participants) | 23
  Lesional skin: After 10 STS: Day 57 | -35.6 (23.2)
  Lesional skin: After 10 STS: Day 85: number analyzed (Participants) | 21
  Lesional skin: After 10 STS: Day 85 | -36.2 (21.3)
  Lesional skin: After 10 STS: Week 16: number analyzed (Participants) | 20
  Lesional skin: After 10 STS: Week 16 | -41.2 (20.4)
  Lesional skin: After 15 STS: Day 15: number analyzed (Participants) | 9
  Lesional skin: After 15 STS: Day 15 | -13.3 (23.9)
  Lesional skin: After 15 STS: Day 29: number analyzed (Participants) | 10
  Lesional skin: After 15 STS: Day 29 | -27.0 (16.3)
  Lesional skin: After 15 STS: Day 57: number analyzed (Participants) | 8
  Lesional skin: After 15 STS: Day 57 | -31.4 (22.1)
  Lesional skin: After 15 STS: Day 85: number analyzed (Participants) | 7
  Lesional skin: After 15 STS: Day 85 | -33.7 (18.1)
  Lesional skin: After 15 STS: Week 16: number analyzed (Participants) | 7
  Lesional skin: After 15 STS: Week 16 | -43.1 (20.6)
  Lesional skin: After 20 STS: Day 15: number analyzed (Participants) | 9
  Lesional skin: After 20 STS: Day 15 | -13.6 (26.3)
  Lesional skin: After 20 STS: Day 29: number analyzed (Participants) | 10
  Lesional skin: After 20 STS: Day 29 | -25.5 (16.1)
  Lesional skin: After 20 STS: Day 57: number analyzed (Participants) | 9
  Lesional skin: After 20 STS: Day 57 | -33.3 (23.4)
  Lesional skin: After 20 STS: Day 85: number analyzed (Participants) | 7
  Lesional skin: After 20 STS: Day 85 | -32.2 (22.5)
  Lesional skin: After 20 STS: Week 16: number analyzed (Participants) | 7
  Lesional skin: After 20 STS: Week 16 | -42.6 (22.1)
  Non-Lesional skin: After 5 STS: Day 15: number analyzed (Participants) | 24
  Non-Lesional skin: After 5 STS: Day 15 | 8.2 (22.1)
  Non-Lesional skin: After 5 STS: Day 29: number analyzed (Participants) | 23
  Non-Lesional skin: After 5 STS: Day 29 | -1.0 (10.2)
  Non-Lesional skin: After 5 STS: Day 57: number analyzed (Participants) | 22
  Non-Lesional skin: After 5 STS: Day 57 | 0.2 (14.8)
  Non-Lesional skin: After 5 STS: Day 85: number analyzed (Participants) | 20
  Non-Lesional skin: After 5 STS: Day 85 | 3.4 (18.2)
  Non-Lesional skin: After 5 STS: Week 16: number analyzed (Participants) | 20
  Non-Lesional skin: After 5 STS: Week 16 | -0.8 (13.6)
  Non-Lesional skin: After 10 STS: Day 15: number analyzed (Participants) | 25
  Non-Lesional skin: After 10 STS: Day 15 | 10.6 (29.0)
  Non-Lesional skin: After 10 STS: Day 29: number analyzed (Participants) | 24
  Non-Lesional skin: After 10 STS: Day 29 | -2.6 (14.2)
  Non-Lesional skin: After 10 STS: Day 57: number analyzed (Participants) | 23
  Non-Lesional skin: After 10 STS: Day 57 | -1.8 (18.2)
  Non-Lesional skin: After 10 STS: Day 85: number analyzed (Participants) | 21
  Non-Lesional skin: After 10 STS: Day 85 | 2.4 (24.3)
  Non-Lesional skin: After 10 STS: Week 16: number analyzed (Participants) | 21
  Non-Lesional skin: After 10 STS: Week 16 | -0.5 (17.9)
  Non-Lesional skin: After 15 STS: Day 15: number analyzed (Participants) | 25
  Non-Lesional skin: After 15 STS: Day 15 | 17.7 (37.6)
  Non-Lesional skin: After 15 STS: Day 29: number analyzed (Participants) | 24
  Non-Lesional skin: After 15 STS: Day 29 | -4.8 (20.5)
  Non-Lesional skin: After 15 STS: Day 57: number analyzed (Participants) | 23
  Non-Lesional skin: After 15 STS: Day 57 | -1.2 (25.5)
  Non-Lesional skin: After 15 STS: Day 85: number analyzed (Participants) | 21
  Non-Lesional skin: After 15 STS: Day 85 | 3.8 (31.0)
  Non-Lesional skin: After 15 STS: Week 16: number analyzed (Participants) | 21
  Non-Lesional skin: After 15 STS: Week 16 | -2.0 (23.5)
  Non-Lesional skin: After 20 STS: Day 15: number analyzed (Participants) | 25
  Non-Lesional skin: After 20 STS: Day 15 | 18.6 (37.7)
  Non-Lesional skin: After 20 STS: Day 29: number analyzed (Participants) | 24
  Non-Lesional skin: After 20 STS: Day 29 | -7.5 (25.2)
  Non-Lesional skin: After 20 STS: Day 57: number analyzed (Participants) | 23
  Non-Lesional skin: After 20 STS: Day 57 | -0.8 (27.7)
  Non-Lesional skin: After 20 STS: Day 85: number analyzed (Participants) | 21
  Non-Lesional skin: After 20 STS: Day 85 | 5.5 (38.2)
  Non-Lesional skin: After 20 STS: Week 16: number analyzed (Participants) | 21
  Non-Lesional skin: After 20 STS: Week 16 | -2.1 (26.2)

25. Secondary Outcome: Percent Change From Baseline in TEWL After 5, 10, 15 and 20 STS on Normal Skin in Healthy Volunteers at Day 15, 29, 57, 85 and Week 16
Description: TEWL assessment: a noninvasive in vivo measurement of water loss across stratum corneum that is used to characterize SBF. TEWL combined with STS measures SBF. With STS, uppermost layers of skin are peeled away using adhesive discs. Normal skin areas for TEWL assessment and STS were identified at Baseline ('predefined skin area'). Within predefined normal skin areas, 3 closely adjacent non-overlapping spots identified for subsequent SBF assessment. TEWL was measured prior to STS and after 5, 10, 15 and 20 STS on pre-defined normal skin areas at specified time points. STS assessment was done at Baseline (Week 0, Day 1), Day 57 and Week 16 on 1st spot; at Day 15 on 2nd spot and at Day 29 and Day 85 on 3rd spot. Percent change from Baseline at specified time points in TEWL after STS on normal skin in healthy volunteers were reported in this OM.
Time Frame: Baseline, Day 15, 29, 57, 85 and Week 16
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Healthy Volunteer
Number analyzed (Participants) | 23
percent change
  After 5 STS: Day 15 | 15.9 (27.8)
  After 5 STS: Day 29 | 5.2 (24.5)
  After 5 STS: Day 57 | 16.0 (27.6)
  After 5 STS: Day 85 | 5.8 (26.3)
  After 5 STS: Week 16 | 1.2 (21.9)
  After 10 STS: Day 15: number analyzed (Participants) | 22
  After 10 STS: Day 15 | 17.6 (31.3)
  After 10 STS: Day 29: number analyzed (Participants) | 21
  After 10 STS: Day 29 | 6.8 (27.8)
  After 10 STS: Day 57: number analyzed (Participants) | 22
  After 10 STS: Day 57 | 13.7 (25.9)
  After 10 STS: Day 85: number analyzed (Participants) | 22
  After 10 STS: Day 85 | 3.1 (26.8)
  After 10 STS: Week 16: number analyzed (Participants) | 22
  After 10 STS: Week 16 | -2.0 (23.5)
  After 15 STS: Day 15: number analyzed (Participants) | 21
  After 15 STS: Day 15 | 32.3 (80.8)
  After 15 STS: Day 29: number analyzed (Participants) | 22
  After 15 STS: Day 29 | 1.6 (37.1)
  After 15 STS: Day 57 | 15.3 (49.1)
  After 15 STS: Day 85 | 1.7 (60.2)
  After 15 STS: Week 16 | -7.2 (35.8)
  After 20 STS: Day 15 | 44.2 (107.8)
  After 20 STS: Day 29: number analyzed (Participants) | 22
  After 20 STS: Day 29 | 31.1 (94.8)
  After 20 STS: Day 57 | 22.0 (63.2)
  After 20 STS: Day 85 | 8.5 (89.4)
  After 20 STS: Week 16 | -5.8 (46.0)

26. Secondary Outcome: Absolute Change From Baseline in TEWL After 5, 10, 15 and 20 STS on Normal Skin in Healthy Volunteers at Day 15, 29, 57, 85 and Week 16
Description: TEWL assessment: a noninvasive in vivo measurement of water loss across stratum corneum that is used to characterize SBF. TEWL combined with STS measures SBF. With STS, uppermost layers of skin are peeled away using adhesive discs. Normal skin areas for TEWL assessment and STS were identified at Baseline ('predefined skin area'). Within predefined normal skin areas, 3 closely adjacent non-overlapping spots identified for subsequent SBF assessment. TEWL was measured prior to STS and after 5, 10, 15 and 20 STS on pre-defined normal skin areas at specified time points. STS assessment was done at Baseline (Week 0, Day 1), Day 57 and Week 16 on 1st spot; at Day 15 on 2nd spot and at Day 29 and Day 85 on 3rd spot. Absolute change from Baseline at specified time points in TEWL after STS on normal skin in healthy volunteers were reported in this OM.
Time Frame: Baseline, Day 15, 29, 57, 85 and Week 16
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: grams per square meter per hour
Arm/Group | Healthy Volunteer
Number analyzed (Participants) | 23
grams per square meter per hour
  After 5 STS: Day 15 | 1.7 (3.8)
  After 5 STS: Day 29 | 0.2 (2.9)
  After 5 STS: Day 57 | 1.6 (4.2)
  After 5 STS: Day 85 | 0.1 (3.3)
  After 5 STS: Week 16 | 0.0 (2.7)
  After 10 STS: Day 15: number analyzed (Participants) | 22
  After 10 STS: Day 15 | 2.1 (5.5)
  After 10 STS: Day 29: number analyzed (Participants) | 21
  After 10 STS: Day 29 | 0.4 (4.0)
  After 10 STS: Day 57: number analyzed (Participants) | 22
  After 10 STS: Day 57 | 1.5 (5.4)
  After 10 STS: Day 85: number analyzed (Participants) | 22
  After 10 STS: Day 85 | -0.4 (4.2)
  After 10 STS: Week 16: number analyzed (Participants) | 22
  After 10 STS: Week 16 | -0.8 (4.0)
  After 15 STS: Day 15: number analyzed (Participants) | 21
  After 15 STS: Day 15 | 3.3 (15.0)
  After 15 STS: Day 29: number analyzed (Participants) | 22
  After 15 STS: Day 29 | -1.9 (8.8)
  After 15 STS: Day 57 | 0.5 (12.8)
  After 15 STS: Day 85 | -3.0 (12.7)
  After 15 STS: Week 16 | -4.5 (11.1)
  After 20 STS: Day 15 | 5.6 (22.4)
  After 20 STS: Day 29: number analyzed (Participants) | 22
  After 20 STS: Day 29 | 1.9 (20.5)
  After 20 STS: Day 57 | 0.0 (19.7)
  After 20 STS: Day 85 | -5.2 (23.3)
  After 20 STS: Week 16 | -8.0 (19.2)

27. Secondary Outcome: Percent Change From Baseline in Area Under the Curve (AUC) of TEWL on Lesional and Non-lesional Skin in AD Patients at Day 15, 29, 57, 85 and Week 16
Description: TEWL assessment: a noninvasive in vivo measurement of water loss across stratum corneum that is used to characterize SBF. TEWL combined with STS measures SBF. TEWL AUC done over defined number of STS was used to reflect the overall integrity of the stratum corneum. LS and non-LS areas for TEWL assessment and STS was identified at Baseline ('predefined skin area'). Within the predefined LS and non-LS areas, 3 closely adjacent non-overlapping spots identified for subsequent SBF assessment (3 spots on LS, 3 spots on non-LS). TEWL was measured prior to STS and after 5, 10, 15 and 20 STS on pre-defined LS and non-LS areas at specified time points. TEWL AUC was a composite measure before and after 5, 10, 15 and 20 STS at each specified time point. AUC of TEWL: calculated for each visit using trapezoidal rule. Percent change from Baseline at specified time points in TEWL AUC in AD participants were reported in this OM.
Time Frame: Baseline, Day 15, 29, 57, 85 and Week 16
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Atopic Dermatitis Patients
Number analyzed (Participants) | 26
percent change
  Lesional skin: Day 15: number analyzed (Participants) | 25
  Lesional skin: Day 15 | -17.0 (37.5)
  Lesional skin: Day 29: number analyzed (Participants) | 24
  Lesional skin: Day 29 | -20.5 (39.3)
  Lesional skin: Day 57: number analyzed (Participants) | 23
  Lesional skin: Day 57 | -24.3 (49.2)
  Lesional skin: Day 85: number analyzed (Participants) | 21
  Lesional skin: Day 85 | -24.5 (56.9)
  Lesional skin: Week 16: number analyzed (Participants) | 21
  Lesional skin: Week 16 | -29.2 (43.5)
  Non-Lesional skin: Day 15: number analyzed (Participants) | 25
  Non-Lesional skin: Day 15 | 52.4 (99.9)
  Non-Lesional skin: Day 29: number analyzed (Participants) | 24
  Non-Lesional skin: Day 29 | 1.0 (48.8)
  Non-Lesional skin: Day 57: number analyzed (Participants) | 23
  Non-Lesional skin: Day 57 | 17.7 (89.4)
  Non-Lesional skin: Day 85: number analyzed (Participants) | 21
  Non-Lesional skin: Day 85 | 29.5 (105.6)
  Non-Lesional skin: Week 16: number analyzed (Participants) | 21
  Non-Lesional skin: Week 16 | 19.4 (97.6)

28. Secondary Outcome: Absolute Change From Baseline in Area Under the Curve of TEWL on Lesional and Non-lesional Skin in AD Patients at Day 15, 29, 57, 85 and Week 16
Description: TEWL assessment: noninvasive in vivo measurement of water loss across stratum corneum, used to characterize SBF. TEWL combined with STS measures SBF. TEWL AUC done over defined number of STS was used to reflect overall integrity of the stratum corneum. LS and non-LS areas for TEWL assessment and STS was identified at Baseline ('predefined skin area'). Within predefined LS and non-LS areas, 3 closely adjacent non-overlapping spots identified for subsequent SBF assessment (3 spots on LS, 3 spots on non-LS). TEWL was measured prior to STS and after 5,10,15 and 20 STS on pre-defined LS and non-LS areas at specified time points. TEWL AUC was a composite measure before and after 5, 10, 15 and 20 STS at each specified time point. AUC of TEWL: calculated for each visit using trapezoidal rule. Absolute change from Baseline at specified time points in TEWL AUC in AD participants were reported in this OM. Expanded unit of measure is number of skin tape stripping*grams per square meter per hour.
Time Frame: Baseline, Day 15, 29, 57, 85 and Week 16
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: nsts*g/m^2/hour
Arm/Group | Atopic Dermatitis Patients
Number analyzed (Participants) | 26
nsts*g/m^2/hour
  Lesional skin: Day 15: number analyzed (Participants) | 25
  Lesional skin: Day 15 | -229.6 (400.8)
  Lesional skin: Day 29: number analyzed (Participants) | 24
  Lesional skin: Day 29 | -278.0 (384.1)
  Lesional skin: Day 57: number analyzed (Participants) | 23
  Lesional skin: Day 57 | -292.3 (409.2)
  Lesional skin: Day 85: number analyzed (Participants) | 21
  Lesional skin: Day 85 | -284.8 (448.7)
  Lesional skin: Week 16: number analyzed (Participants) | 21
  Lesional skin: Week 16 | -321.2 (464.2)
  Non-Lesional skin: Day 15: number analyzed (Participants) | 25
  Non-Lesional skin: Day 15 | 230.9 (536.0)
  Non-Lesional skin: Day 29: number analyzed (Participants) | 24
  Non-Lesional skin: Day 29 | -66.2 (299.3)
  Non-Lesional skin: Day 57: number analyzed (Participants) | 23
  Non-Lesional skin: Day 57 | -22.4 (380.9)
  Non-Lesional skin: Day 85: number analyzed (Participants) | 21
  Non-Lesional skin: Day 85 | 59.1 (483.9)
  Non-Lesional skin: Week 16: number analyzed (Participants) | 21
  Non-Lesional skin: Week 16 | -27.7 (348.1)

29. Secondary Outcome: Percent Change From Baseline in Area Under the Curve of TEWL on Normal Skin in Healthy Volunteers at Day 15, 29, 57, 85 and Week 16
Description: TEWL assessment: a noninvasive in vivo measurement of water loss across stratum corneum that is used to characterize SBF. TEWL combined with STS measures SBF. TEWL AUC done over defined number of STS was used to reflect the overall integrity of the stratum corneum. Normal skin areas for TEWL assessment and STS was identified at Baseline ('predefined skin area'). Within the predefined normal skin areas, 3 closely adjacent non-overlapping spots identified for subsequent SBF assessment. TEWL measured prior to STS and after 5,10,15 and 20 STS on pre-defined normal skin areas at specified time points. TEWL AUC was a composite measure before and after 5, 10, 15 and 20 STS at each specified time point. AUC of TEWL: calculated for each visit using trapezoidal rule. Percent Change from Baseline at specified time points in TEWL AUC in healthy volunteers were reported in this OM.
Time Frame: Baseline, Day 15, 29, 57, 85 and Week 16
Population: Analyzed on mITT population. Here, overall number of participants analyzed = participants evaluable for this OM. Data for this OM was not planned to be collected and analyzed for Atopic Dermatitis Patients arm as pre-specified in the protocol.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Healthy Volunteer
Number analyzed (Participants) | 23
percent change
  Day 15 | 23.3 (51.2)
  Day 29 | 2.6 (39.6)
  Day 57 | 14.0 (36.2)
  Day 85 | 1.0 (45.6)
  Week 16 | -5.5 (30.5)

30. Secondary Outcome: Absolute Change From Baseline in TEWL Area Under the Curve (AUC) on Normal Skin in Healthy Volunteers at Day 15, 29, 57, 85 and Week 16
Description: TEWL assessment: a noninvasive in vivo measurement of water loss across stratum corneum that is used to characterize SBF. TEWL combined with STS measures SBF. TEWL AUC done over defined number of STS was used to reflect the overall integrity of the stratum corneum. Normal skin areas for TEWL assessment and STS was identified at Baseline ('predefined skin area'). Within the predefined normal skin areas, 3 closely adjacent non-overlapping spots identified for subsequent SBF assessment. TEWL measured prior to STS and after 5,10,15 and 20 STS on pre-defined normal skin areas at specified time points. TEWL AUC was a composite measure before and after 5, 10, 15 and 20 STS at each specified time point. AUC of TEWL: calculated for each visit using trapezoidal rule. Absolute change from Baseline at specified time points in TEWL AUC in healthy volunteers were reported in this OM. Expanded unit of measure is number of skin tape stripping*grams per square meter per hour.
Time Frame: Baseline, Day 15, 29, 57, 85 and Week 16
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: nsts*g/m^2/hour
Arm/Group | Healthy Volunteer
Number analyzed (Participants) | 23
nsts*g/m^2/hour
  Day 15 | 49.6 (157.9)
  Day 29 | -17.7 (133.2)
  Day 57 | 20.9 (145.2)
  Day 85 | -31.2 (148.4)
  Week 16 | -46.5 (125.5)

ADVERSE EVENTS:
Time Frame: For AD participants: from first dose (i.e., Day 1) of IMP administration up to end of treatment visit (i.e., Day 113). For healthy volunteers: from signature of consent form to end of study (i.e., from screening to Day 141).
Description: Reported adverse events (AEs) and deaths were treatment-emergent AEs (TEAEs) that occurred, worsened or became serious during TEAE period of AD participants (defined as time from 1st IMP administration to end of treatment) and for healthy volunteers: from signature of consent form to end of study. Analysis was performed on safety population.
Arm/Group | Healthy Volunteer | Atopic Dermatitis Patients
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 13/26 | 20/26
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Volunteer (N=26) | Atopic Dermatitis Patients (N=26)
Dental Restoration Failure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foreign Body In Eye (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Limb Injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Blood Pressure Abnormal (Investigations) | 1 (1) | 0 (0)
Conjunctivitis Allergic (Eye disorders) | 0 (0) | 1 (1)
Dry Eye (Eye disorders) | 0 (0) | 1 (1)
Noninfective Conjunctivitis (Eye disorders) | 0 (0) | 2 (2)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Food Poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis Atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin Burning Sensation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Abscess Limb (Infections and infestations) | 0 (0) | 1 (1)
Covid-19 (Infections and infestations) | 1 (1) | 0 (0)
Herpes Zoster (Infections and infestations) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1)
Tooth Abscess (Infections and infestations) | 1 (1) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Food Allergy (Immune system disorders) | 0 (0) | 2 (2)
Injection Site Reaction (General disorders) | 0 (0) | 5 (6)
Medical Device Site Erythema (General disorders) | 1 (1) | 0 (0)
Medical Device Site Haemorrhage (General disorders) | 2 (2) | 2 (2)
Medical Device Site Pain (General disorders) | 1 (1) | 0 (0)
Medical Device Site Urticaria (General disorders) | 1 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Breast Tenderness (Reproductive system and breast disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2020-07-28): https://cdn.clinicaltrials.gov/large-docs/17/NCT04447417/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-06): https://cdn.clinicaltrials.gov/large-docs/17/NCT04447417/SAP_001.pdf